CLINICAL TRIAL: NCT05584891
Title: Comparative Study Between Radical Mastoidectomy With and Without Mastoid Obliteration Operations in Pediatric Population
Brief Title: Radical Mastoidectomy Versus Mastoid Oblitration in Pediatric Population
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Michael Abdo, principal investigator, Assiut University
Other Study IDs: mariambarkat
Record Dates: First submitted 2022-10-14; First posted 2022-10-18 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Paediatric Cholesteatoma
MeSH Terms: interventions — Mastoidectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group 1: radical mastoidectomy
  Interventions: Procedure: mastoidectomy and mastoid oblitration
- group2: mastoid obliteration operation.
  Interventions: Procedure: mastoidectomy and mastoid oblitration

INTERVENTIONS:
Procedure: mastoidectomy and mastoid oblitration — Forty pediatric patients with cholesteatoma indicated for radical mastoidectomy or modified radical mastoidectomies will be enrolled in our study and we will be grouped into two groups: one will undergo radical mastoidectomy alone and their operation results will be compared to other group which includes twenty pediatric patients with mastoid obliteration operation.

SUMMARY:
Chronic otitis media (COM) has a significant impact on health issues since prehistoric time. It is a global disease, seen in all the continents of world having different environmental and socioeconomic background. COM is characterized as a permanent abnormality of the pars tensa or flaccida, most likely a result of earlier acute otitis media, negative middle ear pressure or otitis media with effusion. COM squamous active (cholesteatoma) is a type of COM, which is a mass formed by keratinizing squamous epithelium in the middle ear and/or mastoid, subepithelial connective tissue and by the progressive accumulation of keratin debris with/without surrounding inflammatory reaction.

DETAILED DESCRIPTION:
Paediatric cholesteatoma spread more extensively through the temporal bone than in adult as the temporal bone in children is well pneumatized. The disease in children is frequently more extensive and expanding, with more involvement of the peri-labyrinthine cells and petrous apex. It is a commonly encountered disease entity which requires prompt surgical management as early as possible. The management of cholesteatoma is solely surgical.

Comparatively the pediatric population has higher rates of recurrent and residual disease, possibly due to anatomic and physiologic differences. Eustachian tube anatomy and dysfunction predisposes children to more frequent infections and retraction pockets. Thus posing a greater challenge than in adults in treating cholesteatom.

The goals of surgery are to eliminate epithelial and bone disease thoroughly and prevent the recurrence, produce a dry and safe ear and to restore serviceable hearing

ELIGIBILITY:
Inclusion Criteria:

- 1. Patient suffering from chronic suppurative otitis media, attico-antral (squamous) disease.

2. Age less than or equal to 18 years.

Exclusion Criteria:

- 1. Patient having an intracranial complication of chronic suppurative otitis media.

2. Bony erosion of sinus plate or dural plate or bone covering the Trautmann's triangle with granulations over the erosion in patients undergoing mastoid obliteration operation.

Ages: 2 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: peadeatric population
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-06-30 (Estimated); Primary Completion 2024-08-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
best option for cholestatoma | about 3 years
  what operation with least recurrence

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university hospital, Asyut, Egypt

REFERENCES:
- [Result] Alves RD, Cabral Junior F, Fonseca AC, Bento RF. Mastoid Obliteration with Autologous Bone in Mastoidectomy Canal Wall Down Surgery: a Literature Overview. Int Arch Otorhinolaryngol. 2016 Jan;20(1):76-83. doi: 10.1055/s-0035-1563382. Epub 2015 Aug 24. PMID 26722350